CLINICAL TRIAL: NCT04673201
Title: Viscotrabeculotomy Versus Trabeculectomy With "MMC" for the Management of Medically Uncontrolled Steroid Induced Glaucoma
Brief Title: Management Steroid Induced Glaucoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amr Mohammed Elsayed Abdelkader, Lecturer of ophthalmology, Mansoura University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R.20.11.1083 - 2020/11/20
Record Dates: First submitted 2020-12-12; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Steroid-Induced Glaucoma
Keywords: Steroid induced glaucoma; Trabeculectomy; Trabeculotomy; MMC

STUDY DESIGN:
Intervention Model Description: Retrospective comparative study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Viscotrabeculotomy group (Active Comparator): Management of medically uncontrolled steroid induced glaucoma by viscotrabeculomy technique
  Interventions: Procedure: Viscotrabeculotomy Versus trabeculectomy with "MMC"
- Trabeculectomy with "MMC" group (Active Comparator): Management of medically uncontrolled steroid induced glaucoma by trabeculotomy with MMC
  Interventions: Procedure: Viscotrabeculotomy Versus trabeculectomy with "MMC"

INTERVENTIONS:
Procedure: Viscotrabeculotomy Versus trabeculectomy with "MMC" — Viscotrabeculotomy involved the creation of a partial thickness scleral flap, followed by localization of Schlemm's canal by radial incisions.High viscosity sodium hyaluronate was injected into Schlemm's canal.Trabeculotomy was completed using the standard metal Harm's trabeculotome.The scleral flap was then secured and conjunctival closure ensued.Trabeculectomy technique involved a creation of a limbal-based conjunctival flap, followed by creation of a half-thickness sclera flap. MMC was applied underneath the conjunctival flap.The procedure was completed with both sclera and conjunctiva closed by 10/0 nylon sutures.

SUMMARY:
Purpose:

To assess the safety and efficacy of Viscotrabeculotomy Versus trabeculectomy with MMC for the management of medically uncontrolled steroid induced glaucoma.

Patients and methods:

A retrospective review of 86 eyes of 67 patients with medically uncontrolled SIG who underwent either viscotrabeculotomy (VT) or trabeculectomy with MMC (Trab-MMC) at Mansoura Ophthalmic Center (Mansoura, Egypt) between January 2008, and December 2017 was conducted.

Keywords:

Steroid induced glaucoma, trabeculectomy, trabeculotomy and MMC.

DETAILED DESCRIPTION:
Introduction:

Steroid induced glaucoma(SIG) is a form of open-angle glaucoma associated with various modalities of corticosteroid administration such as oral, intravenous, inhaled, ocular instilled, intravitreal, and periocular u.Some histologic studies have reported the accumulation of extracellular matrices including basement membrane-like material, fine fibrillar-like material or proteoglycans in the trabecular meshwork (TM) of SIG patients. These observations suggest that such accumulation could lead to an increased resistance to aqueous outflow in the TM of SIG patients.Surgical procedures for intraocular pressure (IOP) reduction in eyes with SIG include trabeculectomy, trabeculotomy,viscocanalostomy and laser trabeculoplasty. Although several case series have shown that these surgeries are effective for IOP reduction, surgical outcomes for SIG are not fully understood due to lack of large case-control studies aiming to investigate the success rates of trabeculotomy in SIG eyes.It has previously been reported that trabeculotomy more effectively reduces IOP in adult Japanese patients with exfoliative glaucoma than in primary open-angle glaucoma (POAG).This IOP lowering effect in eyes with exfoliative glaucoma is thought to be attributable to the relief of abnormally increased outflow resistance that was induced by the accumulation of exfoliative material within the TM. For the same reason, trabeculotomy has been the surgical procedure of choice for adult patients with SIG among Japanese surgeons.Honjo etal previously showed that trabeculotomy helped to reduce IOPs to 21 mm Hg or less in 14 Japanese patients with SIG. However, some questions still without answers for example, whether trabeculotomy with its modifications for SIG offers better IOP management than other surgeries such as trabeculectomy with mitomycin C (MMC), or which characteristics of patients with SIG show better prognosis after trabeculotomy. Therefore the purpose of this retrospective study was to compare the long term surgical outcomes of viscotrabeculectomy(VT) and trabeculectomy with mitomycin C (Trab-MMC) in patients with uncontrolled steroid induced glaucoma.

Subjects and methods:

A retrospective review of 86 eyes of 67 patients with medically uncontrolled SIG who underwent either viscotrabeculotomy (VT) or trabeculectomy with MMC (Trab-MMC) at Mansoura Ophthalmic Center (Mansoura, Egypt) between January 2008, and December 2017 was conducted. The research conformed to the provisions of the Declaration of Helsinki. The confidentiality of the data was ensured. The VT group included 45 eyes and the Trab-ologen group included 41 eyes.

Demographic and clinical data were retrieved from the records such as age at surgery, gender, best-corrected visual acuity (BCVA, LogMAR), intraocular pressure (IOP), gonioscopy, number of glaucoma medications, surgical details and postoperative complications. Steroid-induced glaucoma eyes were defined as open-angle eyes with an IOP elevation of 22 mm Hg or more after the administration of corticosteroid. Glaucoma surgery was performed when IOP was persistently elevated despite maximal tolerated IOP-lowering therapy with potential or actual compromise of optic nerve structure (progressive optic nerve cupping) and/or function (deterioration of visual field testing). All patients were required to sign informed consent forms before surgery.

Viscotrabeculotomy (VT) performed in this study involved the creation of a partial thickness (about 50% thickness) quadrangular (4x4 mm) scleral flap, followed by localization of Schlemm's canal by radial incisions straddling the limbus. High viscosity sodium hyaluronate (Healon GV, Pfizer, NY, USA) was then slowly injected into both ends of Schlemm's canal. Trabeculotomy was completed using the standard metal Harm's trabeculotome (Geuder Instruments, Heidelberg, Germany). Rotation of these probes achieved 120-degree opening of the trabecular meshwork. Next, a small amount of sodium hyaluronate was injected through the open ends of the canal of Schlemm and along the trabeculotomy openings. The scleral flap was then secured tightly with interrupted 10/0 Nylon sutures and conjunctival closure ensued.

Trabeculectomy technique involved a creation of a limbal-based conjunctival flap, followed by creation of a 3 x 4 rectangular half-thickness sclera flap. MMC was applied in a concentration of 0.03% for 3 minutes through soaked surgical sponge inserted underneath the conjunctival flap and spread of a large surface area posterior to the limbus and planned scleral flap site then thoroughly irrigated by 200mL of sterile normal saline. The procedure was completed in the usual manner with both sclera and conjunctiva closed by 10/0 nylon sutures. Postoperative treatment for both groups consisted of topical steroids (dexamethasone) and antibiotic (ofloxacin) five times a day with gradual taper over a period of 5 weeks.

Surgical success was defined at the end of the 4 years of follow up as an IOP between 6 and 21 mmHg and /or IOP reduction greater than 35 % of baseline throughout the entire follow-up period. Absolute success was defined as success being achieved without medications, and qualified success was defined as achieving success with adjunctive medications. Failure was defined as not meeting the above criteria, or any return to the operating theatre for glaucoma reoperation, or loss of vision to no light perception or hypotony (IOP <6 mmHg on 2 occasions after 3 months from the operation). A minimum follow-up of 3 years was required for inclusion in the study.

During the follow up period, eyes that were labelled as "Failure" at any follow up time point were excluded from the data analysis from that follow up time point to the end of the study period (48 months). Follow up was maintained to the patient as part of the patient care service routinely provided by the study setting. The patients' postoperative data was collected from records at day 1, week 1, month 1, month 3, month 6, month 12, month 18, month 24, month 30, month 36 and month 48.

ELIGIBILITY:
Inclusion Criteria:

* Eyes with steroid induced glaucoma when IOP was persistently elevated despite maximal tolerated IOP-lowering therapy with potential or actual compromise of optic nerve structure (progressive optic nerve cupping) and/or function (deterioration of visual field testing)
* A minimum follow-up of 3 years was required for inclusion in the study

Exclusion Criteria:

* Oher causes and types of glaucoma

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2020-11-21 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Absolute success | 4 years
  an IOP between 6 and 21 mmHg and /or IOP reduction greater than 35 % of baseline throughout the entire follow-up period without medications,
qualified success | 4 years
  an IOP between 6 and 21 mmHg and /or IOP reduction greater than 35 % of baseline throughout the entire follow-up period with medications,
Failure | 4 years
  not meeting the above criteria, or any return to the operating theatre for glaucoma reoperation, or loss of vision to no light perception or hypotony (IOP <6 mmHg on 2 occasions after 3 months from the operation)

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university ophthalmic center, Al Mansurah, Dakahlyia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code